CLINICAL TRIAL: NCT06085547
Title: Rural Tailored COVID-19 Communication and SARS-CoV-2 Antibody Testing Evaluation and Uptake
Brief Title: Rural Tailored COVID-19 Communication to Promote SARS-CoV-2 Antibody Testing in Saliva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Johns Hopkins University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Todd Lucas, C.S. Mott Endowed Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 00005016; U01CA260469 (NIH)
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: SARS-CoV2 Infection
Keywords: SARS-CoV-2; COVID-19; Rural Health Disparities; Health Communication; Rural Health; Antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study will use a two-group design (Video tutorial: general versus rural-targeted). Half of White rural participants will receive general video education/messaging and half of White rural participants will be assigned to an intervention condition that includes rural-targeted information about SARS-CoV-2 antibody testing.
Who Masked: Participant
Masking Description: Participants will be unaware of their assignment to a general versus rural-targeted condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White Rural: General (Active Comparator): White rural participants receive "general consumption" video information about SARS-CoV-2 antibody testing.
  Interventions: Behavioral: General SARS-CoV-2 Communication
- White Rural: Rural-Targeted (Experimental): White rural participants receive rural-targeted video information about SARS-CoV-2 antibody testing.
  Interventions: Behavioral: Rural-Targeted SARS-CoV-2 Communication

INTERVENTIONS:
Behavioral: General SARS-CoV-2 Communication — SARS-CoV-2 video tutorial is for general consumption and does not include rural-targeted information
  Arms: White Rural: General
Behavioral: Rural-Targeted SARS-CoV-2 Communication — SARS-CoV-2 video tutorial includes a two and a half minute video based messaging adjunct meant to enact a rural-targeted framing of health information presented to White rural individuals.
  Arms: White Rural: Rural-Targeted

SUMMARY:
This study seeks to evaluate communication strategies for better encouraging understanding and uptake of salivary SARS-CoV-2 antibody testing among individuals residing in rural Northern Michigan. This iteration will consider individuals recruited from rural Northern Michigan and assess individuals' willingness to participate in home-based saliva sample collections.

DETAILED DESCRIPTION:
Rural Americans are at higher risk of many severe COVID-19 related health outcomes. These disparities are likely to endure given lower vaccination uptake in many rural communities, and also the continued emergence of SARS-COV-2 variants, even as overall vaccination rates and COVID-19 treatments improve. Better understanding and addressing rural disparities in COVID-19 could be aided by SARS-CoV-2 antibody testing that can measure herd immunity, assess vaccination efficacy and uptake, and perhaps inform re-vaccination strategies. However, implementing antibody testing education and outreach in rural contexts poses unique challenges, including that many rural communities remain skeptical of COVID-19 testing and treatment. Moreover, rural communities are racially and regionally diverse, including predominantly White populations in some rural regions, but largely African American in others. Such diversity highlights that tailoring the use of specific antibody communication strategies to particular rural contexts is critical. Another challenge posed by rural contexts is in implementing biological sample collections, including effectively distributing and receiving biospecimen collection kits and ensuring proper sample collections. Taken together, there is an urgent need to develop and evaluate communication and collection strategies that can better promote SARS-CoV-2 antibody testing in diverse rural contexts. This study seeks to evaluate communication strategies for better encouraging understanding and uptake of salivary SARS-CoV-2 antibody testing among individuals residing in rural Northern Michigan. The central hypothesis is that rural Americans will be receptive to antibody testing when communication is specifically tailored, and when non-invasive home-based salivary collection is used. The rationale is that combining effective rural health communication with home-based salivary testing will reduce skepticism and mistrust, and promote uptake that can lead to better grasping and addressing rural disparities in COVID-19. The clinical trial aims for this study are to 1) develop and compare the effects of tailored rural videos about antibody testing to general antibody education videos on salivary antibody testing attitudes, intentions, and behavior among rural White Americans residing in Michigan, and rural African Americans residing in Arkansas; 2) compare effects of tailored rural videos on activation of medical mistrust among rural White Americans in Michigan and rural African Americans in Arkansas when considering antibody testing; and 3) develop, evaluate, and compare the efficacy and fidelity of a protocol for home-based salivary collection in rural contexts that includes sending, collecting, receiving and successfully assaying for SARS-CoV-2 antibodies using salivary collection kits. In this study iteration, the investigators will consider individuals recruited from rural Northern Michigan and assess individuals' willingness to participate in home-based saliva sample collections.

ELIGIBILITY:
Inclusion Criteria:

* White, 18 or older

Exclusion Criteria:

* All who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Flint Journal Building, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available per requirements and sharing structures established by NCI "SeroNet" initiative.
Supporting Information: Analytic Code
Time Frame: Upon Study Completion

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 264 enrolled participants, 207 met inclusion criteria and were randomized to a video group. Of the 207 participants who participated in the survey, 13 participants were filtered out for inattentiveness.
Period: Overall Study
Arm/Group | White Rural: General | White Rural: Rural-Targeted
Started | 100 | 94
Completed | 100 | 94
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | White Rural: General | White Rural: Rural-Targeted | Total
Number analyzed (Participants) | 100 | 94 | 194
Age, Customized [Count of Participants; unit: Participants]
  18-21 years | 0 | 0 | 0
  22-40 years | 47 | 43 | 90
  >= 41 | 53 | 51 | 104
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 147
  Male | 26 | 21 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 100 | 94 | 194
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 100 | 94 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number (Percentage) of Participants Requested to Participate in Home-based Saliva-based SARS-CoV-2 Antibody Testing.
Description: Number (percentage) of participants who respond "yes" to be included in the offer to participate in no cost home-based SARS-CoV-2 salivary antibody testing.
Time Frame: Immediately following didactic study portion and health communication randomization on day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | White Rural: General | White Rural: Rural-Targeted
Number analyzed (Participants) | 100 | 94
Participants | 91 | 88

2. Primary Outcome: Number (Percentage) of Participants Who Completed Home-based Salivary Antibody Testing.
Description: Number (Percentage) of participants that requested to participate in antibody testing who actually complete antibody testing.
Time Frame: 8 weeks from the day of consenting to participate in the home-based salivary-based SARS-CoV-2 antibody testing.
Measure: Count of Participants; unit: Participants
Arm/Group | White Rural: General | White Rural: Rural-Targeted
Number analyzed (Participants) | 91 | 88
Participants | 77 | 70

3. Primary Outcome: Theory of Planned Behavior Antibody Testing Outcomes
Description: Self-report measures of antibody testing attitudes, norms, perceived control, and intentions to be screened are each adapted from published research (Lucas et al., 2021). These items are constructed following recommended procedures to ensure construct validity and adequate behavioral specificity (Fishbein & Ajzen, 2011). All items use Likert-type scales that range from 1 (Strongly Agree) to 7 (Strongly Disagree).
Time Frame: collected immediately, up to 1 hour
Measure: Mean (Standard Deviation); unit: Units on a Scale (Minimum:1, Maximum:7)
Arm/Group | White Rural: General | White Rural: Rural-Targeted
Number analyzed (Participants) | 100 | 94
Units on a Scale (Minimum:1, Maximum:7)
  SARS-CoV-2 Antibody Testing Attitudes | 5.97 (.966) | 5.97 (.910)
  SARS-CoV-2 Antibody Testing Normative Beliefs | 4.01 (1.244) | 3.85 (1.158)
  Antibody Testing Perceived Behavioral Control | 6.06 (1.026) | 6.02 (1.092)
  Antibody Testing Intentions | 4.80 (1.487) | 4.92 (1.455)

4. Primary Outcome: Antibody Testing Rural-Adapted Anticipatory Racism
Description: Extent to which participants believe that rural racism-related factors would diminish the value of SARS-CoV-2 antibody testing for self (Seven-point Likert rating, with higher scores indicating greater Anticipatory Racism).
Time Frame: Immediately following didactic study portion and health communication randomization on day 1.
Population: All participants for whom Rural-adapted Anticipatory Racism measure was successfully recorded immediately following messaging randomization.
Measure: Mean (Standard Deviation); unit: Units on a Scale (Minimum:1, Maximum:7)
Arm/Group | White Rural: General | White Rural: Rural-Targeted
Number analyzed (Participants) | 100 | 94
Units on a Scale (Minimum:1, Maximum:7) | 1.63 (.885) | 2.18 (1.166)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | White Rural: General | White Rural: Rural-Targeted
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/94
Other Adverse Events (participants affected / at risk) | 0/100 | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT06085547/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT06085547/SAP_001.pdf